CLINICAL TRIAL: NCT00056316
Title: Reducing Depression in Dementia Caregivers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Missouri, St. Louis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Ann M. Steffen, Ph.D./Associate Professor of Psychology, University of Missouri-St. Louis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21MH061956 (NIH); R21MH061956 (NIH); DSIR AT-GS
Record Dates: First submitted 2003-03-10; First posted 2003-03-11 (Estimated); Results first posted 2008-11-19 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Depression
Keywords: Caregiving; Dementia; Alzheimer's; Depression; Technology; Treatment
MeSH Terms: conditions — Depression; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Skills Training (Experimental): Multicomponent behavioral intervention using 10-session video series (Steffen, et al., 2001) workbook (Steffen, et al., 2001), and weekly telephone coaching sessions.
  Interventions: Behavioral: Behavioral Skills Training: Experimental
- Basic Education (Active Comparator): Participants receive 37-page Basic Care Guide (Education Institute, 2001) and bi-weekly telephone calls by a trained staff member.
  Interventions: Behavioral: Basic Education

INTERVENTIONS:
Behavioral: Basic Education — Participants receive 37-page Basic Care Guide (Education Institute, 2001) and bi-weekly telephone calls by a trained staff member.
  Arms: Basic Education
Behavioral: Behavioral Skills Training: Experimental — Multicomponent behavioral intervention using 10-session video series (Steffen, et al., 2001) workbook (Steffen, et al., 2001), and weekly telephone coaching sessions.
  Arms: Behavioral Skills Training

SUMMARY:
The purpose of this study was to develop and examine the initial impact of a distance-based intervention for female family dementia caregivers. As stated in the original proposal, the primary hypothesis of the study was that family caregivers who participated in the Video Intervention would show greater reduction in psychological distress (i.e., on measures of depression and emotional distress following problematic patient behaviors) compared to those in the Basic Education condition, and that this effect would be maintained over time (3 and 6 months post-tx).

DETAILED DESCRIPTION:
Family caregivers of individuals with dementia commonly report depressive symptoms, along with other forms of emotional distress. This study compared the effectiveness of two home-based interventions to reduce levels of depressed, anxious, and other negative moods in women living with a family member with dementia. Eligible caregivers were randomly assigned to participate in either a video/workbook/telephone coaching intervention, or to a basic education condition consisting of a workbook and supportive telephone calls. Participants were evaluated for psychosocial distress after treatment, and at 3- and 6-months following the end of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver and dementia pt live in the same home
* Resident of following states: Il,IN, IO, KS, MI, MN, MO, NB,WI

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2002-01; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Steffen, PhD, Principal Investigator — University of Missouri, St. Louis
Locations (1):
- University of Missouri-St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Steffen AM. Anger management for dementia caregivers: A preliminary study using video and telephone interventions. Behavior Therapy 31:281-299, 2000.
- [Background] Steffen AM, McKibbin C, Zeiss AM, Gallagher-Thompson D, Bandura A. The revised scale for caregiving self-efficacy: reliability and validity studies. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P74-86. doi: 10.1093/geronb/57.1.p74. PMID 11773226
- [Derived] Gonzalez-Fraile E, Ballesteros J, Rueda JR, Santos-Zorrozua B, Sola I, McCleery J. Remotely delivered information, training and support for informal caregivers of people with dementia. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD006440. doi: 10.1002/14651858.CD006440.pub3. PMID 33417236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from 10/2001 to 3/2004. Project information was distributed to Alzheimers Association Chapters and Area Agencies on Aging (AAA's) in Midwestern USA (IO, IL,IN, KS, MI, MO, MN, NB,WI).
Pre-assignment Details: All enrolled participants who completed consent procedures were randomly assigned to groups.
Period: Overall Study
Arm/Group | Behavioral Skills Training | Basic Education
Started | 33 | 41 (over-enrolled due to potential higher rates of drop-out.)
Completed | 30 | 38
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death/NH placement of pt | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Skills Training | Basic Education | Total
Number analyzed (Participants) | 33 | 41 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 10 | 15 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (11.9) | 62.9 (9.6) | 61.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 41 | 74
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 41 | 74

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory II (Beck, Steer & Brown, 1996)
Description: 21-item self-report instrument to assess severity of symptoms of depression. There is a four-point scale for each item ranging from 0 to 3. The total continuous score can range from 0 to 63 points, with higher scores reflective of greater severity.
Time Frame: Pre-intervention intake assessment, conducted 7-14 days prior to start of intervention
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Behavioral Skills Training | Basic Education
Number analyzed (Participants) | 33 | 41
Points on a scale | 14.27 (8.07) | 16.93 (8.46)

2. Secondary Outcome: Negative Affect Schedule (Watson, Clark & Tellegen, 1988)
Description: 10 item self-report assessment of negative affects. Participants rate items on a scale from 1 to 5, based on the strength of emotion where 1 = "very slightly or not at all," and 5 = "extremely". The total continuous score may range from 10 to 50, with higher values indicative of stronger negative emotion.
Time Frame: Pre-intervention intake assessment, conducted 7-14 days prior to start of intervention
Population: All participants who were randomized into the study were included in the analyses (i.e., Intention to treat). Missing values were replaced with the Last Observation Carried Forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Behavioral Skills Training | Basic Education
Number analyzed (Participants) | 33 | 41
Points on a scale | 24.15 (6.72) | 24.17 (7.25)

3. Primary Outcome: Primary Outcome: Beck Depression Inventory II (Beck, Steer & Brown, 1996)
Description: as for outcome 1
Time Frame: Post-intervention, assessed 4-14 days after final intervention session.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Behavioral Skills Training | Basic Education
Number analyzed (Participants) | 33 | 41
Points on a scale | 10.25 (7.23) | 13.83 (8.36)
Statistical Analysis 1: Comparison: Behavioral Skills Training vs Basic Education; Test type: Superiority or Other; p = .05, t-test, 2 sided; Mean Difference (Final Values) = 1.93 — Mean difference is equal to Behavioral Skills Intervention minus Basic Education Control

4. Secondary Outcome: Secondary Outcome: Negative Affect Scale (Watson, Clark & Tellegen, 1988)
Description: as for outcome 2
Time Frame: Post-intervention, assessed 4-14 days after final intervention session.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Behavioral Skills Training | Basic Education
Number analyzed (Participants) | 33 | 41
Points on a scale | 18.52 (5.66) | 21.63 (6.99)
Statistical Analysis 1: Comparison: Behavioral Skills Training vs Basic Education; Test type: Superiority or Other; p = .05, t-test, 2 sided; Mean Difference (Final Values) = 2.07 — Mean difference is equal to Behavioral Skills Intervention minus Basic Education Control

ADVERSE EVENTS:
Arm/Group | Behavioral Skills Training | Basic Education
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No